CLINICAL TRIAL: NCT03512470
Title: A Clinical Study, Spontaneous, Randomized and Controlled, on the Prevention of Surgical Wound Complications for Aneurysmal Thoracoabdominal Aortic Disease by Using the "PREVENA ™" Negative Topical Pressure System (TVAC STUDY)
Brief Title: Clinical Study on the Prevention of Surgical Wound Complications for Aneurysmal Thoracic-abdominal Aortic Pathology Using the "PREVENA" System
Acronym: TVAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Baccellieri Domenico, Principal Investigator, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17/INT/2018
Record Dates: First submitted 2018-04-19; First posted 2018-04-30 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Toraco Abdominal Aneurysm
Keywords: surgical wound; Prevena System
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sistema Prevena ™ (TVAC) (Experimental): Negative topical pressure system (Sistema Prevena ™).
  Interventions: Device: Sistema Prevena ™(TVAC)
- Standard medication (Active Comparator): Standard medication with sterile gauzes and a TNT patch or medicated patch
  Interventions: Other: Standard medication

INTERVENTIONS:
Device: Sistema Prevena ™(TVAC) — The medications with a negative topical pressure system (Sistema Prevena ™) will be applied directly in the Operating Room. Thereafter medication will be checked in the inpatient ward after 48 h from the intervention, evaluating the possible absorption of exudate on the surface. If no absorption are detected within 48 hours, the medication won't be removed and renewed in the 7th day (± 2 days) post-operative; and to follow every 7 (± 2 days) until the points are removed. If the wound continues to progress towards recovery, the protocol will continue until discharge and / or rehabilitation and / or surgery.
  Arms: Sistema Prevena ™ (TVAC)
Other: Standard medication — standard medication in use (sterile gauze and TNT patch or medicated patches).
  Arms: Standard medication

SUMMARY:
The patients will be randomized into two groups of 100 subjects each one. One arm will be randomized to treatment with a negative topical pressure system (Sistema Prevena ™); while the other arm ("control group") will be randomized to treatment with standard medication with sterile gauzes and a TNT patch or medicated patch as normal traditional medication in use.

The medications with a negative topical pressure system (Sistema Prevena ™) will be applied directly in the Operating Room. Thereafter the medication will be checked in the inpatient ward after 48 hours from the intervention, evaluating the possible absorption of exudate on the surface. If no absorption are detected within 48 hours, the medication won't be removed. The medication will be renewed in the 7th day (± 2 days) post-operative; and to follow every 7 (± 2 days) until the points are removed. If the wound continues to progress towards recovery, the protocol will continue until discharge and / or rehabilitation and / or surgery. For each evaluation the photograph of the medication must be taken (which will be deprived of all the identifying elements of the patient).

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years;
* patients of any sex, race, age, who have accepted to participate in the study by signing the informed consent form of the study.
* patients with surgical wounds to treat thoracic-abdominal aortic pathology.

Exclusion Criteria:

* patients with established sepsis;
* patients with septic recurrence;
* patients with sensitivity to silver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Reduction of surgical site infections | 14 days after surgery
  Decrease in the percentage of surgical site infections and / or surgical wound dehiscence within 14 days of surgery

SECONDARY OUTCOMES:
Reduction of adverse events | 12 month
  decrease in the percentage of surgical reoperation
Reduction of adverse events | 12 month
  decrease in the percentage of seromas / hematomas

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cutting KF, White RJ. Criteria for identifying wound infection--revisited. Ostomy Wound Manage. 2005 Jan;51(1):28-34. PMID 15695833
- [Background] Matatov T, Reddy KN, Doucet LD, Zhao CX, Zhang WW. Experience with a new negative pressure incision management system in prevention of groin wound infection in vascular surgery patients. J Vasc Surg. 2013 Mar;57(3):791-5. doi: 10.1016/j.jvs.2012.09.037. Epub 2013 Jan 9. PMID 23312938
- [Derived] Cristino MA, Nakano LC, Vasconcelos V, Correia RM, Flumignan RL. Prevention of infection in aortic or aortoiliac peripheral arterial reconstruction. Cochrane Database Syst Rev. 2025 Apr 22;4(4):CD015192. doi: 10.1002/14651858.CD015192.pub2. PMID 40260835